CLINICAL TRIAL: NCT03253302
Title: Laparoscopic Assisted transAnal Total Mesorectal Excision for Rectal cAncer in Low Site :A Prospective,Multi-center, Patients Registry Trial in China (LATERAL Trial)
Brief Title: Laparoscopic Assisted Transanal Total Mesorectal Excision for Rectal Cancer in Low Site
Acronym: LATERAL-01
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Ruijin Hospital (Other); The First Hospital of Jilin University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, assistant dean, professor, Beijing Friendship Hospital
Other Study IDs: CR-TaTME
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Rectal Cancer
Keywords: transanal surgery; total mesorectal excision; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present, surgical resection is still the main treatment for the potential cure of rectal cancer. Total mesorectal excision (TME) is the gold standard. The traditional laparoscopic or open surgery for some special patients is really difficult, especially for male, prostate hypertrophy, obesity, low tumor and pelvic stenosis patients to expose the gap around the mesorectum and separate to the pelvic floor. While transanal total mesorectal excision (TaTME) approach could be more directly separate the low mesorectum and relatively simple to complete distal rectal transection, which would bring some considerable advantages. Although active learning from abroad, laparoscopic assisted TaTME surgery is now in its infancy in China. It is urgent for clinical studies to obtain the results in China. This multicenter, observational study will help to encourage research in this field and to obtain data on the safety and efficacy of this procedure in Chinese patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the rectum by biopsy
* the lower edge of the tumor from the anal margin less than 10cm according to MRI or rigid endoscopy
* tumor diameter less than 4cm
* baseline clinical stage I-III: cT1-3 N0-2 M0 (AJCC v7)
* tolerable to surgery
* be able to understand and willing to participate in this trial with signature

Exclusion Criteria:

* history of malignant colorectal neoplasia
* recent diagnosis with other malignancies
* patients requiring emergency surgery such as obstruction，perforation and bleeding
* tumor involving adjacent organs, anal sphincter, or levator ani muscle
* muti-focal colorectal cancer
* preoperative poor anal function, anal stenosis, anal injury, or fecal incontinence
* history of inflammatory bowel disease or familial adenomatous polyposis
* participating in other clinical trails
* can not tolerate the surgery
* history of serious mental illness
* pregnancy or lactating women
* preoperative uncontrolled infection
* the researchers believe the patients should not enrolled in

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lower rectal cancer patients who are suitable and willing to accept laparoscopy- assisted TME procedure and also agree with the trial
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Positive rate of circumferential resection margin (CRM) of the specimens | 10 days after surgery
  Circumferential resection margin (CRM) is the distance between the deepest point of tumor in the primary cancer and the margin of resection in the retroperitoneum or mesentery by pathological examination. CRM 0-1mm is defined as positive, while >1mm is negative.

SECONDARY OUTCOMES:
The grade score of the specimens integrity | 10 days after surgery
  shows the quality of the specimens: grade 1 is bad gross specimen which means incomplete mesorectum and pelvic fascia, and muscle layer can be see >5mm; grade 3 is high quality gross specimen, which means the specimen is cylindrical, mesorectum and pelvic fascia are complete; grade 2 is between 1and 3.
The distance between lower tumor margin and the lower reaction margin | 10 days after surgery
  shows the oncological safety of the surgery by pathological examination. Reports should contain the distance between lower tumor margin and the lower reaction margin.
local recurrence rate | 3 years after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the operative time | 30 days after surgery
  preoperative safety containing operation information, complication information.
postoperative hospital stay | 3 year after surgery
  recovery information.
the score of postoperative life | 6 months after surgery
  quality of life contains two scales: Wexner scale and EORTC QLQ-CR29 scale, which show quality of life and the anal function.
disease free survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
overall survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the rate of postoperative complications | 30 days after surgery
  preoperative safety containing operation information, complication information.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China